CLINICAL TRIAL: NCT05315167
Title: A Phase 1/2, Open-label Study Evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Prime Efficacy of PRJ1-3024 in Subjects with Advanced Solid Tumors
Brief Title: A Phase I/II Study to Evaluate the Safety, Pharmacokinetics and Efficacy of PRJ1-3024 in Subjects with Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zhuhai Yufan Biotechnologies Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PRJ1-3024-001; CXHL2101725 (Other: CDE)
Record Dates: First submitted 2022-03-29; First posted 2022-04-07 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-10

CONDITIONS: Advanced Solid Tumor; Advanced Solid Malignancies
Keywords: Maximum tolerated dose; Recommended Phase 2 dose; Dose Escalation; Hematopoietic progenitor kinase 1; PRJ1-3024
MeSH Terms: conditions — Hereditary Sensory and Autonomic Neuropathies

STUDY DESIGN:
Intervention Model Description: Part 1 is a Phase 1, open label, 3+3 dose escalation study to determine the safety and preliminary efficacy of PRJ1-3024. Upon completing Phase 1 and depending on data obtained, dose expansion may proceed in Phase 2 to confirm the tolerability and efficacy of the RP2D of PRJ1-3024 .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Monotherapy Escalation (Experimental): 3+3 Dose escalation arm with PRJ1-3024 which will begin with 2 subjects treated at the lowest planned dose level. PRJ1-3024 is administered orally once daily. The starting dose is 80mg/day.
  Interventions: Drug: PRJ1-3024
- Monotherapy Exploration of the recommended dose (Experimental): Upon completing Phase 1 and depending on data obtained, dose expansion may proceed in Phase 2 with several cohorts enrolled to confirm the tolerability of the RP2D of PRJ1-3024 (determined in Phase 1). PRJ1-3024 is administered orally once daily. The starting dose is determined by clinical effecacy data from Phase 1, and treatment may continue for up to 2 years as long as the subject experiences clinical benefit in the opinion of the Investigator and shows no signs or symptoms of unequivocal progression of disease.
  Interventions: Drug: PRJ1-3024

INTERVENTIONS:
Drug: PRJ1-3024 — PRJ1-3024 is provided as capsules and is administered orally once a day.

SUMMARY:
This is a multicenter, open-label study to assess the safety and preliminary efficacy and to determine the maximum tolerated dose (MTD) or maximum administration dose (MAD) and recommended Phase 2 doses (RP2D) of PRJ1-3024 in subjects with relapsed/refractory solid tumors. The study consists of two parts, one is a 3+3 dose escalation study and another is a pharmaceutical extension of RP2D.

DETAILED DESCRIPTION:
Using dose escalation, the study will evaluate the safety, tolerability, PK, and pharmacodynamics of PRJ1-3024 and will determine the maximum tolerated dose in subjects with advanced solid tumors.

Participants with advanced solid tumor will receive PRJ1-3024 daily as an oral therapy and test the impact of of PRJ1-3024 on tumors.

This study will find the safe and tolerable recommended dose in subjects with advanced solid tumors in a open-label, 3+3 dose escalation study and use the RP2D to assess the preliminary efficacy of PRJ1-3024 in a long-term extension study.

ELIGIBILITY:
- Key Inclusion Criteria:

* Histologically or cytologically confirmed locally advanced (unresectable) or metastatic r/r solid tumors for which no standard therapy is available or for whom standard therapy is considered unsuitable or intolerable.
* Male or non-pregnant, non-lactating female subjects age ≥18 years.
* ECOG Performance Status 0~1.
* Has at least 1 measurable lesion as defined by RECIST 1.1 criteria .
* Life expectancy of >3 months, in the opinion of the Investigator.
* Able to take oral medications and willing to record daily adherence to investigational product.
* Adequate hematologic parameters unless clearly due to the disease under study.
* Adequate renal and hepatic function
* Able to understand and willing to sign a written informed consent form.

Key Exclusion Criteria:

* History of another malignancy
* Known symptomatic brain metastases requiring >10 mg/day of prednisolone.
* Significant cardiovascular disease.
* Known active HBV, HCV, AIDS-related illness.
* Has received a live vaccine within 30 days.
* History of active autoimmune disorders, or ongoing immunosuppressive therapy or ongoing .
* Continuance of toxicities due to prior radiotherapy or chemotherapy agents that do not recover to < Grade 2.
* Receiving concurrent anti-cancer therapy, investigational product, strong inhibitors or inducers of cytochrome P450 3A (CYP3A) .
* Prior treatment with hematopoietic progenitor kinase 1 (HPK1) inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Estimated)
Dates: Start 2022-05-30 (Actual); Primary Completion 2027-05-15 (Estimated); Study Completion 2027-11-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicity (DLT) events during the DLT monitoring period | Day 1 to Day 21
  Safety listings and pharmacokinetic listings will be used for evaluation

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | 24 months
  Characterized by type, seriousness, relationship to study treatment, timing, and severity.
Pharmacokinetic parameter# Accumulation ratio | 24 months
  to estimate the accumulation of PRJ1-3024 from time 0 to the time of last quantifiable concentration after multiple administration
Objective response rate (ORR) | 24 months
  estimated by the proportion of subjects having a complete response (CR) or partial response (PR) with use of RECIST v1.1 criteria.
Duration of response (DOR) | 24 months
  defined as time from the first occurrence of a documented objective response to the time of relapse or death from any cause.
Pharmacokinetic parameter#AUC0-last# | 24 months
  Area under the concentration-time curve AUC from time 0 to the time of the last quantifiable concentration
Pharmacokinetic parameter#Maximum observed concentration (Cmax) | 24 months
  assessed as time from time 0 to the time of the last quantifiable concentration

CONTACTS AND LOCATIONS:
Overall Officials: Hui ouyang, Dr., Study Director — VP
Locations (5):
- China (5):
  - The first affiliated hospital of Zhengzhou University, Zhengzhou, Henan
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Cancer hospital of the University of Chinese Academy of Sciences, Hangzhou, Zhejiang
  - Beijing Cancer Hospital, Beijing
  - The Fifth Medical Center of PLA General Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No